CLINICAL TRIAL: NCT01363960
Title: Retinopathy of Prematurity:Summary of a Decade
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Murat KÜÇÜKEVCİLİOĞLU, MD, Gulhane Military Medical School
Other Study IDs: Retinopathy of prematurity
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Retinopathy of Prematurity
Keywords: Incidence; neonatal care; retinopathy of prematurity; risk factors
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neonates with retinopathy of prematurity: all neonates meet the criteria:
  1. a BW of less than 1501 gram (g)
  2. born at a GA of 34 weeks (wk) or less and
  3. selected infants with an unstable clinical course were included

SUMMARY:
The aim of the study is to evaluate our 10 year experience of retinopathy of prematurity screening.

ELIGIBILITY:
Inclusion Criteria:

* Neonates either with a BW of less than 1501 gram (g) or born at a GA of 34 weeks (wk) or less
* selected infants with an unstable clinical course were included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neonates with Retinopathy of of prematurity
Sampling Method: Probability Sample
Enrollment: 609 (Actual)
Dates: Start 1999-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of neonates developed retinopathy of prematurity | ten years
risk factors contributing to ROP development | ten years
  mechanic ventilation. oxygen therapy, respiratory distress syndrome, sepsis, intraventricular, hemorrhage, blood transfusion v.s

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Military Medical School Training Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: retinopathy of prematurity — http://www.ncbi.nlm.nih.gov/pubmed